CLINICAL TRIAL: NCT03198325
Title: Monitored Antiretroviral Pause in Chronic HIV-Infected Subjects With Long-Lasting Suppressed Viremia (APACHE Study)
Brief Title: Monitored Antiretroviral Pause in Chronic HIV-Infected Subjects With Long-Lasting Suppressed Viremia
Acronym: APACHE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS San Raffaele (Other)
Responsible Party: Principal Investigator, Castagna Antonella, Professor, Ospedale San Raffaele
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: APACHE Study
Record Dates: First submitted 2017-06-21; First posted 2017-06-26 (Actual); Last update posted 2024-02-09 (Actual); Status verified 2024-02

CONDITIONS: HIV Seropositivity
Keywords: HIV-1
MeSH Terms: conditions — HIV Seropositivity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Interruption of antiretroviral therapy (Experimental): Patients willing to stop antiretroviral therapy will stop ART.The occurrence of two consecutive HIV-1 RNA values >50 copies/mL or the occurrence of stage B or C AIDS-defining events will be criteria for ART resumption or any serious non-AIDS clinical event at least potentially related to treatment interruption.
  Interventions: Other: Stop of ART

INTERVENTIONS:
Other: Stop of ART — Patients willing to stop antiretroviral therapy will stop ART.The occurrence of two consecutive HIV-1 RNA values >50 copies/mL or the occurrence of stage B or C AIDS-defining events will be criteria for ART resumption or any serious non-AIDS clinical event at least potentially related to treatment interruption.

SUMMARY:
Prospective, open-label, single arm, non-randomized, proof-of-concept study. Eligible patients will sign a written informed consent and will be followed-up at screening, baseline (ART interruption) and at 1, 2, 3, 4, 6, 8, 10, 12, 16, 24, 32, 40, 48 weeks thereafter or at ART resumption.

The study visits will include: general clinical assessment, routine laboratory tests including: creatinine, phosphorus, calcium, alkaline phosphatase, AST, ALT, fasting glucose, total cholesterol, HDL- and LDL-cholesterol, triglycerides, CD4+ cell count and CD4+/CD8+ ratio.

Additional 30 mL of peripheral blood will be withdrawn at study visits for further virological, and immunological investigations and for bio-banking purposes.

During follow-up, the occurrence of two consecutive HIV-1 RNA values >50 copies/mL or the occurrence of stage B or C AIDS-defining events or any serious non-AIDS clinical event at least potentially related to treatment interruption will be criteria for ART resumption.

All patients with HIV-RNA<50 copies/mL at week 48 (end of the study) will resume their baseline ART regimen.

The main demographic, clinical and therapy information will be accurately recorded at the study visits in an electronic Case Report Form.

DETAILED DESCRIPTION:
The aim of this proof-of-concept study on adult (>18 and <65 years old), chronically HIV-1 infected individuals with undetectable viremia for ≥10 years, undetectable HIV-DNA, CD4+≥500 cells/µL and no evidence of detectable residual viremia for ≥5 years is to evaluate the frequency of spontaneous control of virus replication after ART pausing for up to 12 months and to identify the virological and immunological markers associated with spontaneous control of viral replication.

Prospective, open-label, single arm, non-randomized, proof-of-concept study.

Eligible patients will sign a written informed consent and will be followed-up at screening, baseline (ART interruption) and at 1, 2, 3, 4, 6, 8, 10, 12, 16, 24, 32, 40, 48 weeks thereafter or at ART resumption.

The clinical assessment (study visit) will include: the evaluation of CDC stage, height, weight, systolic and diastolic blood pressure and smoking status, routine laboratory tests [including creatinine, phosphorus, calcium, alkaline phosphatase, AST, ALT, fasting glucose, total cholesterol, HDL- and LDL-cholesterol, triglycerides, CD4+ cell count and CD4+/CD8+ ratio, urine analysis].

Additional 30 mL of peripheral blood will be withdrawn at study visits and stored in a biobank for further investigations.

During follow-up, the occurrence of two consecutive HIV-1 RNA values >50 copies/mL or the occurrence of stage B or C AIDS-defining events will be criteria for ART resumption or any serious non-AIDS clinical event at least potentially related to treatment interruption.

All patients with HIV-RNA<50 copies/mL at week 48 (end of the study) will resume their baseline ART regimen.

The main demographic, clinical and therapy information will be accurately recorded at the study visits in an electronic Case Report Form (eCRF).

ELIGIBILITY:
Inclusion Criteria:

The study will include HIV-1 infected:

* men and non-pregnant women,
* ≥18 and <65 years-old,
* asking to stop therapy,
* with HIV-1 RNA<50 copies/mL for ≥10 years,
* current CD4+≥500 cells/µL,
* HIV-DNA<100 copies/106PBMCs,
* no evidence of detectable residual viremia for ≥5 years .

Exclusion Criteria:

The study will exclude HIV-1 infected subjects:

* significant risk of HIV transmission during IMAP (including evidence of not adopting effective contraception methods and women who wish to be pregnant) in the opinion of the investigator,
* pregnancy and breastfeeding,
* a documented pre-ART HIV-1 RNA<200 copies/mL,
* reactive Hepatitis B virus (HBV) surface antigen,
* positive HCV-RNA at the time of screening,
* current AIDS defining event as defined in category C of the 'Centers for disease control and prevention (CDC)' clinical classification,
* previous diagnosis of diabetes,
* a previous diagnosis of cancer or major adverse cardiac events (MACE) and currently receiving chemotherapy or immuno-modulating agents at the time of screening,
* history of HIV-related thrombocytopenia,
* active renal disease defined as a glomerular filtration rate (calculated by MDRD equation) below 50 mL/min or the presence of HIV associated nephropathy in the past medical history,
* any condition, including psychiatric or psychological disorders that might interfere with adherence to study requirements or safety of the participant,
* prior use of any HIV vaccine and/or non-established experimental therapy,
* active drug or alcohol use or dependence that, in the opinion of the site investigator, would interfere with adherence to study requirements.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2016-07-27 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2018-04 (Actual)

PRIMARY OUTCOMES:
Patients who will not resume antiretroviral regimen | 12 month
  Cumulative proportion of patients who will not resume ART 12 months after IMAP (Monitored Antiretroviral Pause) due to the occurrence of two consecutive HIV-1 RNA values >50 copies/mL or the occurrence of stage B or C AIDS-defining events or any serious non-AIDS clinical event at least potentially related to treatment interruption.

SECONDARY OUTCOMES:
Change in plasma viremia | 1, 2, 3, 4, 6, 8, 10, 12, 16, 24, 32, 40, 48 weeks thereafter or at ART resumption.
  Change in plasma viremia
Change in plasma HIV-DNA | 1, 2, 3, 4, 6, 8, 10, 12, 16, 24, 32, 40, 48 weeks thereafter or at ART resumption.
  Change in plasma HIV-DNA
Change in CD4+ | 1, 2, 3, 4, 6, 8, 10, 12, 16, 24, 32, 40, 48 weeks thereafter or at ART resumption.
  Change in CD4+
Change in CD4+/CD8+ ratio | 1, 2, 3, 4, 6, 8, 10, 12, 16, 24, 32, 40, 48 weeks thereafter or at ART resumption.
  Change in CD4+/CD8+ ratio
Change in virological biomarkers | 1, 2, 3, 4, 6, 8, 10, 12, 16, 24, 32, 40, 48 weeks thereafter or at ART resumption.
  Change in virological biomarkers prior to ART interruption and/or at ART resumption
Change in immunological biomarkers | 1, 2, 3, 4, 6, 8, 10, 12, 16, 24, 32, 40, 48 weeks thereafter or at ART resumption.
  Change in immunological biomarkers prior to ART interruption and/or at ART resumption

CONTACTS AND LOCATIONS:
Locations (1):
- Ospedale San Raffaele Scientific Institute, Milan, Italy

IPD SHARING:
Plan to Share IPD: Yes
Congress and scientific pubblications

REFERENCES:
- [Background] Pau AK, George JM. Antiretroviral therapy: current drugs. Infect Dis Clin North Am. 2014 Sep;28(3):371-402. doi: 10.1016/j.idc.2014.06.001. PMID 25151562
- [Background] Strategies for Management of Antiretroviral Therapy (SMART) Study Group; El-Sadr WM, Lundgren J, Neaton JD, Gordin F, Abrams D, Arduino RC, Babiker A, Burman W, Clumeck N, Cohen CJ, Cohn D, Cooper D, Darbyshire J, Emery S, Fatkenheuer G, Gazzard B, Grund B, Hoy J, Klingman K, Losso M, Markowitz N, Neuhaus J, Phillips A, Rappoport C. CD4+ count-guided interruption of antiretroviral treatment. N Engl J Med. 2006 Nov 30;355(22):2283-96. doi: 10.1056/NEJMoa062360. PMID 17135583
- [Background] Strategies for Management of Antiretroviral Therapy (SMART) Study Group; Emery S, Neuhaus JA, Phillips AN, Babiker A, Cohen CJ, Gatell JM, Girard PM, Grund B, Law M, Losso MH, Palfreeman A, Wood R. Major clinical outcomes in antiretroviral therapy (ART)-naive participants and in those not receiving ART at baseline in the SMART study. J Infect Dis. 2008 Apr 15;197(8):1133-44. doi: 10.1086/586713. PMID 18476292
- [Background] Skiest DJ, Krambrink A, Su Z, Robertson KR, Margolis DM; A5170 Study Team. Improved measures of quality of life, lipid profile, and lipoatrophy after treatment interruption in HIV-infected patients with immune preservation: results of ACTG 5170. J Acquir Immune Defic Syndr. 2008 Dec 1;49(4):377-83. doi: 10.1097/QAI.0b013e31818cde21. PMID 18931631
- [Background] Strategies for Management of Antiretroviral Therapy (SMART) Study Group; Lundgren JD, Babiker A, El-Sadr W, Emery S, Grund B, Neaton JD, Neuhaus J, Phillips AN. Inferior clinical outcome of the CD4+ cell count-guided antiretroviral treatment interruption strategy in the SMART study: role of CD4+ Cell counts and HIV RNA levels during follow-up. J Infect Dis. 2008 Apr 15;197(8):1145-55. doi: 10.1086/529523. PMID 18476293
- [Background] Saez-Cirion A, Bacchus C, Hocqueloux L, Avettand-Fenoel V, Girault I, Lecuroux C, Potard V, Versmisse P, Melard A, Prazuck T, Descours B, Guergnon J, Viard JP, Boufassa F, Lambotte O, Goujard C, Meyer L, Costagliola D, Venet A, Pancino G, Autran B, Rouzioux C; ANRS VISCONTI Study Group. Post-treatment HIV-1 controllers with a long-term virological remission after the interruption of early initiated antiretroviral therapy ANRS VISCONTI Study. PLoS Pathog. 2013 Mar;9(3):e1003211. doi: 10.1371/journal.ppat.1003211. Epub 2013 Mar 14. PMID 23516360
- [Background] Williams JP, Hurst J, Stohr W, Robinson N, Brown H, Fisher M, Kinloch S, Cooper D, Schechter M, Tambussi G, Fidler S, Carrington M, Babiker A, Weber J, Koelsch KK, Kelleher AD, Phillips RE, Frater J; SPARTACTrial Investigators. HIV-1 DNA predicts disease progression and post-treatment virological control. Elife. 2014 Sep 12;3:e03821. doi: 10.7554/eLife.03821. PMID 25217531
- [Background] Ho YC, Shan L, Hosmane NN, Wang J, Laskey SB, Rosenbloom DI, Lai J, Blankson JN, Siliciano JD, Siliciano RF. Replication-competent noninduced proviruses in the latent reservoir increase barrier to HIV-1 cure. Cell. 2013 Oct 24;155(3):540-51. doi: 10.1016/j.cell.2013.09.020. Epub 2013 Oct 24. PMID 24243014
- [Background] Hurst J, Hoffmann M, Pace M, Williams JP, Thornhill J, Hamlyn E, Meyerowitz J, Willberg C, Koelsch KK, Robinson N, Brown H, Fisher M, Kinloch S, Cooper DA, Schechter M, Tambussi G, Fidler S, Babiker A, Weber J, Kelleher AD, Phillips RE, Frater J. Immunological biomarkers predict HIV-1 viral rebound after treatment interruption. Nat Commun. 2015 Oct 9;6:8495. doi: 10.1038/ncomms9495. PMID 26449164
- [Background] Lee SA, Bacchetti P, Chomont N, Fromentin R, Lewin SR, O'Doherty U, Palmer S, Richman DD, Siliciano JD, Yukl SA, Deeks SG, Burbelo PD. Anti-HIV Antibody Responses and the HIV Reservoir Size during Antiretroviral Therapy. PLoS One. 2016 Aug 2;11(8):e0160192. doi: 10.1371/journal.pone.0160192. eCollection 2016. PMID 27483366
- [Background] Siliciano JD, Kajdas J, Finzi D, Quinn TC, Chadwick K, Margolick JB, Kovacs C, Gange SJ, Siliciano RF. Long-term follow-up studies confirm the stability of the latent reservoir for HIV-1 in resting CD4+ T cells. Nat Med. 2003 Jun;9(6):727-8. doi: 10.1038/nm880. Epub 2003 May 18. PMID 12754504
- [Background] Burbelo PD, Lebovitz EE, Notkins AL. Luciferase immunoprecipitation systems for measuring antibodies in autoimmune and infectious diseases. Transl Res. 2015 Feb;165(2):325-35. doi: 10.1016/j.trsl.2014.08.006. Epub 2014 Sep 1. PMID 25241936
- [Background] Assoumou L, Weiss L, Piketty C, Burgard M, Melard A, Girard PM, Rouzioux C, Costagliola D; ANRS 116 SALTO study group. A low HIV-DNA level in peripheral blood mononuclear cells at antiretroviral treatment interruption predicts a higher probability of maintaining viral control. AIDS. 2015 Sep 24;29(15):2003-7. doi: 10.1097/QAD.0000000000000734. PMID 26355572
- [Background] Calin R, Hamimi C, Lambert-Niclot S, Carcelain G, Bellet J, Assoumou L, Tubiana R, Calvez V, Dudoit Y, Costagliola D, Autran B, Katlama C; ULTRASTOP Study Group. Treatment interruption in chronically HIV-infected patients with an ultralow HIV reservoir. AIDS. 2016 Mar 13;30(5):761-9. doi: 10.1097/QAD.0000000000000987. PMID 26730568
- [Background] Cuzin L, Pugliese P, Saune K, Allavena C, Ghosn J, Cottalorda J, Rodallec A, Chaix ML, Fafi-Kremer S, Soulie C, Ouka M, Charpentier C, Bocket L, Mirand A, Guiguet M; Dat'AIDS study group. Levels of intracellular HIV-DNA in patients with suppressive antiretroviral therapy. AIDS. 2015 Aug 24;29(13):1665-71. doi: 10.1097/QAD.0000000000000723. PMID 26372277
- [Background] Zheng L, Bosch RJ, Chan ES, Read S, Kearney M, Margolis DM, Mellors JW, Eron JJ, Gandhi RT; DS Clinical Trials Group (ACTG) A5244 Team. Predictors of residual viraemia in patients on long-term suppressive antiretroviral therapy. Antivir Ther. 2013;18(1):39-43. doi: 10.3851/IMP2323. Epub 2012 Aug 22. PMID 22914318
- [Background] Maggiolo F, Callegaro A, Cologni G, Bernardini C, Velenti D, Gregis G, Quinzan G, Soavi L, Iannotti N, Malfatto E, Leone S. Ultrasensitive assessment of residual low-level HIV viremia in HAART-treated patients and risk of virological failure. J Acquir Immune Defic Syndr. 2012 Aug 15;60(5):473-82. doi: 10.1097/QAI.0b013e3182567a57. PMID 22481602
- [Background] Gianotti N, Canducci F, Galli L, Cossarini F, Salpietro S, Poli A, Nozza S, Spagnuolo V, Clementi M, Sampaolo M, Ceresola ER, Racca S, Lazzarin A, Castagna A. HIV DNA loads, plasma residual viraemia and risk of virological rebound in heavily treated, virologically suppressed HIV-infected patients. Clin Microbiol Infect. 2015 Jan;21(1):103.e7-103.e10. doi: 10.1016/j.cmi.2014.08.004. Epub 2014 Oct 13. PMID 25636935
- [Background] Li JZ, Etemad B, Ahmed H, Aga E, Bosch RJ, Mellors JW, Kuritzkes DR, Lederman MM, Para M, Gandhi RT. The size of the expressed HIV reservoir predicts timing of viral rebound after treatment interruption. AIDS. 2016 Jan 28;30(3):343-53. doi: 10.1097/QAD.0000000000000953. PMID 26588174
- [Background] Tedaldi E, Peters L, Neuhaus J, Puoti M, Rockstroh J, Klein MB, Dore GJ, Mocroft A, Soriano V, Clotet B, Lundgren JD; SMART Study Group and International Network for Strategic Initiatives in Global HIV Trials (INSIGHT). Opportunistic disease and mortality in patients coinfected with hepatitis B or C virus in the strategic management of antiretroviral therapy (SMART) study. Clin Infect Dis. 2008 Dec 1;47(11):1468-75. doi: 10.1086/593102. PMID 18959492
- [Background] Monroe AK, Chander G, Moore RD. Control of medical comorbidities in individuals with HIV. J Acquir Immune Defic Syndr. 2011 Dec 15;58(5):458-62. doi: 10.1097/QAI.0b013e31823801c4. PMID 22083037
- [Derived] Mastrangelo A, Burbelo PD, Galli L, Poli A, Alteri C, Scutari R, Muccini C, Spagnuolo V, Caccia R, Turrini F, Bigoloni A, Galli A, Castagna A, Cinque P. Anti-HIV antibodies are representative of the latent reservoir but do not correlate with viral control in people with long-lasting virological suppression undergoing analytical treatment interruption (APACHE study). J Antimicrob Chemother. 2021 May 12;76(6):1646-1648. doi: 10.1093/jac/dkab060. No abstract available. PMID 33693943